CLINICAL TRIAL: NCT04385121
Title: Psychological Impact of the Hospitalization of a Family Member in Intensive Care for Covid-19 Infection
Acronym: Familles-COVID
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7761
Record Dates: First submitted 2020-04-16; First posted 2020-05-12 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-07

CONDITIONS: Covid-19; Stress Disorders, Post-Traumatic; Anxiety; Depression
Keywords: COVID-19; Psychological impact; Family members
MeSH Terms: conditions — COVID-19; Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnary — Family member's will answer the questionnaires by phone

SUMMARY:
The hospitalization of a patient in intensive care is a traumatic experience for his family members.

With the current COVID-19 epidemic, in view of the high risk of contamination, drastic measures to limit the transmission are necessary, with the creation of spaces dedicated to the care of Covid+ patients, and family are not allowed to visit.

At the Strasbourg University Hospital, visits were prohibited from the start of the epidemic. Information concerning the patient's state of health is therefore delivered to families by telephone, on call by the healthcare team only, every day before 6 p.m. or in the event of a serious event at any time.

The primary purpose of this project is to assess the psychological impact of the hospitalization of a loved one in intensive care for Covid-19 infection at 3 months post-hospitalization, in a context of pandemic with ban on visits.

ELIGIBILITY:
Inclusion Criteria:

* Family member of a Covid-19 positive patient hospitalized in Intensive Care Unit who gave his oral agreement following the communication of the notice of non-opposition.
* A patient is considered to be Covid + if the RT-PCR is positive OR if characteristic images are taken with a chest scanner.
* The family member included in the study is preferably the patient's support person. In the absence of an expression of the patient's will, he is the close referent designated by the family as an interlocutor.

Exclusion Criteria:

* Difficulties in understanding French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Family members of COVID+ patient
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Existence of a post-intensive care syndrome-family ((combined score of the HAD ( Hospital Anxiety and Dépression scale) and IES-R ( Impact of Event Scale-Revised) questionnaires)) | 3 months
  An overall score of 19 or more indicates a major depressive episode (HAD) and a total score of 22 as in favor of significant symptoms of acute stress (IES-R)

CONTACTS AND LOCATIONS:
Overall Officials: Julie HELMS, Principal Investigator — CHU de Strasbourg
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cattelan J, Castellano S, Merdji H, Audusseau J, Claude B, Feuillassier L, Cunat S, Astrie M, Aquin C, Buis G, Gehant E, Granier A, Kercha H, Le Guillou C, Martin G, Roulot K, Meziani F, Putois O, Helms J. Psychological effects of remote-only communication among reference persons of ICU patients during COVID-19 pandemic. J Intensive Care. 2021 Jan 9;9(1):5. doi: 10.1186/s40560-020-00520-w. PMID 33422153